CLINICAL TRIAL: NCT02205021
Title: Compartmental Neck Fat Accumulation and Its Relationship to Cardiovascular Risk and Metabolic Syndrome
Brief Title: Neck Fat Accumulation and Its Relationship to Cardiovascular Risk and Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Torriani, Martin,M.D., Assistant Professor of Radiology, Massachusetts General Hospital
Other Study IDs: 2012P001603
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Accumulation of fat in the neck using tape measures has been linked to increased cardiovascular risk. The investigators' hypothesis is that detailed measures of neck fat using computed tomography will show that specific fat compartments in the neck contribute differently to cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* no history of malignancy at the time of image acquisition
* fasting glucose measured immediately prior to PET/CT

Exclusion Criteria:

* history of neck cancer, radiation therapy, and/or surgery

Ages: 18 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective search of whole-body PET/CT examinations and consecutively selected imaging studies.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Relationship of specific neck compartments to cardiovascular risk | 1 year between PET/CT and cardiometabolic marker measures
  Cardiovascular risk measures were obtained within one year of CT imaging of the neck.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Torriani, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Torriani M, Gill CM, Daley S, Oliveira AL, Azevedo DC, Bredella MA. Compartmental neck fat accumulation and its relation to cardiovascular risk and metabolic syndrome. Am J Clin Nutr. 2014 Nov;100(5):1244-51. doi: 10.3945/ajcn.114.088450. Epub 2014 Sep 3. PMID 25332322